CLINICAL TRIAL: NCT04042883
Title: Acute Normovolemic Hemodilution Using Hydroxyethyl Starch (HES 130/0.4) in Patients Undergoing Off-pump Coronary Artery Bypass Grafting Surgery: Effects on Central and Peripheral Perfusion
Brief Title: Acute Normovolemic Hemodilution in Off-pump CABG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hany Mostafa Esmaeil Osman, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hemodilution off-pump CABG
Record Dates: First submitted 2019-08-01; First posted 2019-08-02 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Acute Normovolemic Hemodilution; Off-Pump Coronary Artery Bypass Surgery
Keywords: Perfusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANH (Active Comparator): 500 ml of blood will be taken from the patient with simultaneous replacement with hydroxyethyl starch (HES 130/0.4) in another IV line
  Interventions: Procedure: Acute normovolemic hemodilution
- Control (No Intervention): No intervention

INTERVENTIONS:
Procedure: Acute normovolemic hemodilution — 500 ml of blood will be taken from the patient with simultaneous replacement with hydroxyethyl starch (HES 130/0.4) in another IV line
  Other Names: ANH
  Arms: ANH

SUMMARY:
To study the effects of Acute normovolemic hemodilution on central and peripheral perfusion in patients Undergoing off-pump coronary artery bypass grafting surgery

DETAILED DESCRIPTION:
Off-pump coronary artery bypass surgery is an alternative to conventional coronary artery bypass grafting using cardiopulmonary bypass (CPB). It avoids adverse effects of CPB such as systemic inflammatory response, impaired myocardial protection, and air or plaque embolism. However, OPCAB surgery involves displacement and manipulation of the heart to expose target coronary arteries. These manipulations cause hemodynamic instability as a result of transient annulo-mitral distortion and acute mitral regurgitation, compression of the right ventricle, and impaired cardiac contractility due to epicardial stabilizers. signs of impaired perfusion such as metabolic acidosis, increased serum lactate and decreased urine output are commonly seen intraoperatively

Excessive surgical bleeding causes hypovolemia and hemodynamic instability, anemia, and reduced oxygen delivery to tissues

Acute normovolemic hemodilution (ANH) is an alternative method of management of intraoperative blood loss, in which a certain volume of blood is collected from the patient, stored at room temperature and replaced by an equal volume of colloid solution. By the end of surgery, this blood is returned to the patient, usually within eight hours of collection, with little deterioration of platelets or coagulation factors

This work aims to study the effects of Acute normovolemic hemodilution on central and peripheral perfusion in patients Undergoing off-pump coronary artery bypass grafting surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for off- pump CABG surgery

Exclusion Criteria:

* Ejection fraction less than 40%
* Hematocrit less than 11 g/dl
* patients with severe renal impairment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-08-10 (Actual); Primary Completion 2020-04-15 (Estimated); Study Completion 2020-04-15 (Estimated)

PRIMARY OUTCOMES:
Central venous oxygen saturation | Intraoperative
  Central venous blood gas analysis
The perfusion index | Intraoperative
  perfusion index derived from pulseoximetry
Serum lactate | Intraoperative
  from arterial blood gas analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt